CLINICAL TRIAL: NCT06278623
Title: Effects of Focal Muscle Vibratory Energy in Patients With Parkinson's Disease: Pilot Prospective Observational Study.
Brief Title: Focal Muscle Vibration in Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4935
Record Dates: First submitted 2023-03-10; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2023-08

CONDITIONS: Parkinson Disease; Postural; Defect; Rehabilitation
MeSH Terms: conditions — Parkinson Disease | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Focal Muscle Vibratory Energy (EVM) Treatment — The patients involved in the study will undergo muscle vibratory stimulation in association with conventional rehabilitation treatment three times a week, for three weeks for a total duration of 9 sessions in association with conventional treatment.
  The vibration will be applied at a frequency of 100 Hz and an amplitude of 0.2 cm for 30 minutes (three sessions of 10 min each with 1 min break in between) three times a week for three weeks at the level of the quadriceps femoris and triceps surae bilaterally for balance improvement and stimulation of proprioception and in the trapezius and trunk extensor muscles bilaterally for pain relief.

SUMMARY:
Postural instability has a major impact on the mobility and daily life activities of Parkinson's disease (PD) patients as it often leads to reduced mobility, insecure stance and falls.

The aim of this study was to evaluate the effect of focal vibration on the static and dynamic balance of a group of Parkinson's disease patients with Hoehn and Yahr (HeY) stage II-III. They underwent three weeks of focal muscle vibration applied to the quadriceps, soles of the feet and trapezius muscles bilaterally in addition to conventional physiotherapy . The static and dynamic balance was assessed at baseline (T0), after 3 weeks of treatment (T1) and after 1 month from the last treatment (T2) with the Tinetti scale and stabilometry evaluations.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a chronic, highly disabling neurodegenerative disorder characterized by bradykinesia, resting tremor, rigidity and postural instability . Postural instability has been shown to have a major impact on the autonomy, mobility and quality of life of these patients as it often leads to insecure stance and falls . Balance control is a complex system involving the integration of vestibular, visual and proprioceptive sensory information. Somatosensory information is derived from a variety of sources, most notably the cutaneous mechanoreceptors in the skin and the muscle spindles . It is well known that a decline in skin sensitivity and proprioceptive input naturally occurs with aging. Moreover, kinesthetic sensory deficits may occur due to systemic and neurologic disorders (e.g., diabetes, stroke etc.). Previous studies have demonstrated that the integration of sensory information is abnormal in PD patients with strong repercussions on motor function, posture, static and dynamic balance and greater reliance on visual input for postural control . The effectiveness of current treatments on postural instability and kinesthetic deficits in PD is controversial. Bartolic et al. observed improvement in postural control after treating rigidity with apomorphine. Wright and colleagues [6] suggest that axial kinesthetic sensitivity worsens with levodopa. Furthermore, important side effects and loss of therapeutic efficacy after years of use of dopaminergic agonists represent a major clinical challenge. Muscle vibration is a safe, non-invasive rehabilitation technique that holds promise for improving mobility and balance in moderate to severe PD patients. It consists of local vibrations applied on selected muscles or tendons by means of a mechanical device.

Stimulation of Ia afferent fibers from muscle spindles and cutaneous receptors strongly increases the exteroceptive and proprioceptive input to the central nervous system (CNS).

This has been shown to induce a plastic modulation of the primary sensory motor cortex andspinal reflexes, with long lasting positive effects on muscle tone and motor control Despite good results obtained in several other neurological conditions, such as post stroke spatial heminattention, spastic hypertonia and motor control impairment , only a few studies exist on the use of focal vibratory energy for posture and gait disorders in Parkinson's disease. Most of the existing experiments in the literature are about whole-body vibration (WBV) which has shown limited efficacy on stability and movement control In contrast, focal vibration applied over the cervical and soleus muscles , and on quadriceps and paraspinal muscles , in conjunction with conventional physiotherapy, has shown positive effects on the patient's balance, risk of falling and quality of gait.

Despite a consistent body of literature on the use of muscle vibration in rehabilitation, there is currently insufficient evidence regarding its application in patients with Parkinson's disease, including muscle targets, duration and frequency of the treatment and technical parameters. Based on these premises, we aimed to evaluate the effects of focal vibration on static and dynamic balance of patients with Parkinson's disease.

This is a prospective, observational, pilot study. Chronic patients with idiopathic Parkinson's disease were recruited from the Physical and Rehabilitation ward of the Agostino Gemelli Foundation University Hospital of Rome.

Each patient underwent focal muscle vibration in association with conventional physiotherapy three times a week, for three weeks, for a total of nine sessions. The vibration wasapplied via a pneumatic vibration device (EVM, Endomedica, Rome, Italy) at a frequenc of 100 Hz and an amplitude of 0.2 mm. Each session consisted of three stimulation trains of 10 min each, interspersed with 1 min of rest. The stimulus was applied at the level of the upper and lower trapezius, quadriceps femoris and sole of the foot bilaterally with the patient in sitting position . The choice of this last target was based on our clinical judgment and recent literature evidence. The feet provide a direct interface between the body and the environment and represent an important sensory structure in the mechanism of postural control. Plantar skin mechanoreceptors transmit crucial information about pressure variations on the sole of the feet which determine reflex postural reactions through activation of antigravitary muscles . Group rehabilitation was carried out after each focal muscle vibration session. Each group consisted of 5 individuals coordinated by an experienced physiotherapist (DR). The physiotherapy program included several exercises according to the literature :

* Exercises for the head and trunk control;
* Strengthening and stabilization of lower limbs and antigravity muscles;
* Stretching of the posterior kinetic chain muscles;
* Exercises aimed at recovering and maintaining a correct posture;
* Coordination and balance exercises;
* Gait training with and without obstacles. Static balance was assessed through a standardized stabilometry exam performed on a "Prokin PK 254 P" device produced by TecnoBody S.r.l. (Dalmine (BG), Italy). The device consists of a static platform (47 cm of circumference) with four piezoelectric sensors positioned at the extremity of the four cardinal points. The temporal resolution was 0.01 s, and the sampling frequency was set at 20 Hz. The patients were asked to stand on the platform for 60 s in a neutral position with the feet forming a 30-degree angle. The test was performed 30" with the eyes open and 30" with the eyes closed. All data were analyzed by the ProKin 36 software in order to calculate the center of pressure (CoP) sway on the X (anterior-posterior) and Y (medio-lateral) axes (mm), the center of pressure (CoP) velocity on the X (anterior-posterior) (AP-vel) and Y (medio-lateral) (ML-Vel) axes (mm/s), the sway path (Perimeter, total length of CoP trajectory (mm) and the area of the ellipse (mm2).

Lower values reflect greater control in maintaining the static balance. We considered as a primary outcome the reduction of the length of adaptive movements in terms of perimeter and sway area as they represent parameters of global stability of the CoP The patients were evaluated at (T0), after 3 weeks of treatment (T1) and after one month from the last treatment session (T2). A Tinetti scale was used to assess the gait and dynamic balance while consecutive stabilometric examinations were performed to assess the static balance. All patients were tested during the "on phase", 45-90 min after the morning dose of levodopa.

The Tinetti scale, also known as performance-oriented mobility assessment (POMA), is a standardized screening modality for gait and balance disorders. It is applied to screen different patient populations including elderly patients and patients with Parkinson's disease. The test assesses a patient's balance and gait using a standardized scoring system comprising 16 items with a maximal score of 28. A score ≤ 18, a score between 19-24 and a score ≥ 25 reflect an overall high, medium and low risk of falls, respectively Numeric rating scale and Mc Gill pain questionaire were used to measure pain at each timing evaluation.

Descriptive analysis was performed using standard procedures for the calculation of frequencies, measure of average position (arithmetic mean) and dispersion indicators.

The differences between pretreatment and post-treatment measures at each timing were analyzed with Student's t-test for paired samples. A p-value < 0.05 for two side test was considered statistically significant. Data analysis was conducted with the software SPSS 1.4

ELIGIBILITY:
Inclusion criteria:

* diagnosis of Parkinson's disease according to the criteria of the Brain Bank of London;
* Hoehn and Yahr stage II-III;
* absence of cognitive impairment
* (MMSE > 24/30); e
* effective pharmacological control of the pathology;
* being part of the PD group-rehabilitation program of our ward for at least one year; -
* acceptance and signature of informed consent.

Exclusion criteria:

* comprised: a diagnosis of atypical Parkinsonism;
* poor pharmacological compensation of the disease;
* diagnosis of other neurological diseases;
* diagnosisof neuromuscular diseases;
* diagnosis of osteo-articular pathologies;
* cognitive impairment (MMSE < 24);
* visual impairment;
* vestibular disorders;
* not being part of our PD group-rehabilitation for at least one year;
* denial of informed consent

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients affected by Parkinson's disease, who refer to the Physiatry clinic of the Gemelli University Hospital Foundation in Rome.
Sampling Method: Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Tinetti scale | Evaluation was performed at (T0), after 3 weeks of treatment (T1) and after one month from the last treatment session (T2)
  balance and deambulation scale. The Tinetti scale, also known as performance-oriented mobility assessment (POMA), It is a standardized screening modality for gait and balance disorders. It is applied to screen different patient populations including elderly patients and patients with Parkinson's disease. The test assesses a patient's balance and gait using a standardized scoring system comprising 16 items with a maximal score of 28. A score ≤ 18, a score between 19-24 and a score ≥ 25 reflect an overall high, medium and low risk of falls, respectively

SECONDARY OUTCOMES:
NRS numeric rating scale of pain | Evaluation was performed at (T0), after 3 weeks of treatment (T1) and after one month from the last treatment session (T2)
  ranges from 0 to 10 with 0 indicating no pain to 10 maximum pain
Stabilometric Test | Evaluation was performed at (T0), after 3 weeks of treatment (T1) and after one month from the last treatment session (T2)
  Static balance evaluation. Static balance was assessed through a standardized stabilometry exam performed on a "Prokin PK 254 P" device produced by TecnoBody S.r.l. (Dalmine (BG), Italy).Data analysed were the center of pressure (CoP) sway on the X (anterior-posterior) and Y (medio-lateral) axes (mm), the center of pressure (CoP) velocity on the X (anterior-posterior) (AP-vel) and Y (medio-lateral) (ML-Vel) axes (mm/s), the sway path (Perimeter, total length of CoP trajectory (mm) and the area of the ellipse (mm2
  ).Lower values reflect greater control in maintaining the static balance.
Mc Gill Pain questionnaire | Evaluation was performed at (T0), after 3 weeks of treatment (T1) and after one month from the last treatment session (T2)
  evaluation of pain. It is composed of 78 words. Respondents choose those that best describe their experience of pain. Scores are tabulated by summing values associated with each word; scores range from 0 (no pain) to 78 (severe pain). Qualitative differences in pain may be reflected in respondent's word choice

CONTACTS AND LOCATIONS:
Overall Officials: gianpaolo ronconi, Principal Investigator — Catholic University of the Sacred Heart
Locations (1):
- Gianpaolo Ronconi, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided